CLINICAL TRIAL: NCT05530538
Title: A Displacement Theory Mobile Health Weight Loss Intervention: A Pilot Clinical Trial
Brief Title: BrainWeighve App Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Children's Hospital Los Angeles (Other); eHealth International, INC. (Unknown)
Responsible Party: Principal Investigator, Vibha Singhal, Principal Investigator, University of California, Los Angeles
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22-1395
Record Dates: First submitted 2022-08-25; First posted 2022-09-07 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-04

CONDITIONS: Weight Loss; Obesity and Overweight
Keywords: Weight Loss; Adolescents; Smartphone App; Obesity; Overweight
MeSH Terms: conditions — Weight Loss; Obesity; Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BrainWeighve Intervention (Experimental): 4-month smartphone-based weight loss intervention for teens based on displacement theory of addictive behaviors
  Interventions: Behavioral: BrainWeighve App

INTERVENTIONS:
Behavioral: BrainWeighve App — 38 total adolescents (14-21 years old) with %BMIp85 will be recruited via various sources (e.g., clinic referrals, flyers, social media advertising) to participate in one of two stages of the study: the beta testing stage or the trial stage. Beta testing will enroll a group of eight teens to test the app for three weeks; participants will be assessed pre- and post-intervention. The app will be modified to incorporate their feedback in order to promote youth engagement. The trial stage will enroll 30 adolescents to participate in a four-month intervention; participants will complete three assessments, baseline, post-intervention (both in-person) and one-month post-intervention (either in-person or virtually).

SUMMARY:
Childhood obesity within the United States has been a growing concern over the past number of years, and if not addressed, leads to detrimental health outcomes for youth as they move into adulthood. The literature suggests that over-eating, especially when framed in terms of food addiction, plays a key role in this epidemic; however, treatment options are time intensive, posing a profound logistical barrier for both the child and parent and often limits or prevents engagement. As research within the field of mHealth has grown, technology-based interventions have gained traction, specifically interactive smartphone applications (apps). Displacement theory, although not new, has been understudied yet provides a strong explanation and treatment plan for addictive type behaviors. The core of this theory posits that problems which one feels they cannot face nor avoid leads to repetitive and irrepressible behaviors; however, if a healthy coping behavior can be learned and utilized, then the unhealthy behavior will cease. The theory lends itself well to being adapted into an mHealth format, making it more easily accessible and more widely used. Grounded in displacement theory, the proposed study aims to develop an app-based weight loss intervention for adolescents with obesity. Information gained regarding the feasibility and acceptability of such an intervention can potentially be replicated and applied to other populations with various addictive behaviors. Helping those with addictive behaviors in a format that has little to no logistical barriers can have a substantial impact on public health. A novel smartphone app will be designed by key stakeholders and refined through the course of the study. 38 total adolescents (14-21 years old) with %BMIp85 will be recruited via various sources (e.g., clinic referrals, flyers, social media advertising) to participate in one of two stages of the study: the beta testing stage or the trial stage. Beta testing will enroll one group of eight teens to test the app for three weeks; participants will be assessed in-person pre- and post-intervention. After each group, the app will be modified to incorporate their feedback in order to promote youth engagement. The trial stage will enroll 30 adolescents to participate in a four-month intervention; participants will complete three assessments, baseline, post-intervention (both in-person) and one-month post-intervention (either in-person or virtually). The study will examine engagement and satisfaction with the app, as well as the intervention's impact on clinical outcome measures (weight and BMI, diet and snacking, and addictive behaviors related to food and substance use) and potential mediators/moderators (motivation for change, perceived stress, and distress tolerance).

DETAILED DESCRIPTION:
Aim 1: To develop a smartphone app aimed at reducing over-eating behaviors among adolescents with obesity based on the theory that addictive behaviors are driven by a displacement mechanism in the brain. Based on displacement theory, over-eating and associated weight gain are the result of situations that individuals feel they cannot successfully face nor avoid. App development will include input from various stakeholders including obesity medicine specialists, pediatric clinicians, psychologists, and individuals living with obesity.

Aim 2: To test and modify the app through an iterative process; one group of 8 teens will beta test the app for three weeks each and provide quantitative and qualitative data used to make changes which facilitate usability and engagement.

Aim 3: Evaluate the feasibility of the app among 30 adolescents (15F;15M) to identify barriers and facilitators to its implementation. We will measure (a) adherence to daily app use with particular focus on the participant's identification of a "Dread List" and the implementation of "Action Plans" aimed at ameliorating stressful situations identified in the list, (b) quantity (#hours per participant) and quality (type and frequency of team member engagement per participant) of support required to promote adherence, (c) satisfaction with the app intervention (qualitative assessment of satisfaction rates, exit interviews, reason for dropouts), and (d) assessment burden. This knowledge will inform the refinement of the intervention for the subsequent larger trial.

Aim 4: Preliminary assessment of the impact of app engagement and usage on clinical outcome measures (weight and BMI, diet and snacking, and addictive behaviors related to food and substance use) and potential mediators/moderators (motivation for change, perceived stress, and distress tolerance).

Hypothesis 1: More engagement with and use of the app will be related to better clinical outcomes; specifically, participants more engaged in the app will show reductions in weight and BMI, over-eating behaviors (self-reported diet recall and snacking), and overall addictive behaviors.

Hypothesis 2: Participants with greater motivation, lower perceived stress, and greater distress tolerance at intake will engage more with the app and have better clinical outcomes; also, those who engage with and use the app more will exhibit increased motivation, lowered perceived stress, and greater distress tolerance which will in turn result in better clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. 14-21 years old
2. Has an iPhone or are willing to use a study iPhone
3. Ability to read and speak English
4. Endorsement of one of the three items listed below on the five-item S-weight questionnaire indicating motivation for change During the last year I haven't done anything to lose weight but I'm planning to do something over the next 30 days.

I've been making an effort to lose weight (by dieting1 and/or exercising2) for less than 6 months.

I've been making an effort to maintain my weight (by dieting1 and/or exercising2) for more than 6 months.

6. Body mass index [BMI] ≥85th percentile for age and gender

Exclusion Criteria:

1. Any psychiatric condition and/or developmental delay which would require immediate or ongoing treatment that would make study participation difficult or harmful
2. Parent/guardian-reported physical, mental of other inability to provide consent or refusal to provide consent for minor children
3. Self-reported diagnosis of Prader-Willi Syndrome, brain tumor, hypothalamic obesity, or other diagnosis associated with obesity
4. Concurrent participation in an alternative weight loss intervention
5. Participation in the study team's previous app weight loss studies (exclusion for trial but not beta testing participants)

Ages: 14 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 38 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Quantity of Engagement with App | 4 months
  Daily engagement as measured by minutes per day each participant spent in the app
Satisfaction with the App as assessed by the Treatment Satisfaction Questionnaire | 4 months
  The TSQ (Cox, Fergus & Swinson, 1994) will be modified and used for this study to provide a quantitative assessment of participant satisfaction with the BrainWeighve app. The measure contains a nine item Likert-scale asking the participant to rate how satisfied they were with the app overall, its ease or difficulty of use, how satisfied they were with the impact the app had on their behaviors and weight loss, and if they would be likely to continue using it outside of a research study.
Quality of Engagement with App | 4 months
  Number of items participant enters over the intervention period for their Dread List and Action Plans

SECONDARY OUTCOMES:
%BMI95 | 5 months
  Weight and height; participants will also be asked to enter their daily weight into the app using their study-provided scale. Adolescents will be instructed to wear minimal clothing during the height and weight measurements. BMI will be calculated as kilograms per meter squared and BMI z-score (zBMI) and excess percent of the 85th percentile (%BMIp85) will be determined utilizing the CDC growth charts (baseline, post-treatment, and 1-month post-treatment.
Automated Self-Administered 24-Hour Dietary Assessment Tool | 5 months
  The ASA-24 is a recall measure developed by the US National Cancer Institute that asks participants to self-report all food and beverages consumed within the past 24-hour period (baseline, post, and 1-month post)
Substance Use as measured by the NIDA Risk Assessment | 5 months
  Substance use will be assessed using items drawn from the NIDA Risk Assessment Questionnaire (1993). This scale asks participants to report past 30-day use of alcohol, marijuana, and "other drugs." (baseline, post, 1-month post)
Perceived Stress Scale | 5 months
  The PSS measures subjective perceptions of distress in one's own life situations on a 10-item, 5-point scale. Based on Lazarus' transactional model of stress and coping, the PSS assesses how well a person feels they can cope with stressors, rather than measuring the nature of the stressors themselves. The measure has demonstrated strong reliability (r > 0.80) and validity in social and health science studies (baseline, post, 1-month post)
Distress Tolerance Scale | 5 months
  The DTS (Simons & Gaher, 2005) is a 15-item self-report measure of ability to withstand emotional distress, measuring four factors: tolerance, appraisal, absorption, and regulation (alpha=.82). (baseline, post, 1-month post)
Mental Health Inventory | 5 months
  One item from the RAND MHI (Veit & Ware, 1983) will be used to provide a general assessment of mental health well-being on a 6-point Likert scale of Extremely Happy to Very Dissatisfied (i.e., "How happy, satisfied, or pleased have you been with your personal life during the past month?"). (baseline, post, 1-month post)
Weight Management Program Diet Questionnaire | 5 months
  A 23-item validated measure used to assess readiness and willingness to make behavioral changes to lose weight. Items are measured on a 5-point Likert scale and are organized into six categories (Goals and Attitudes, Hunger and Eating Cues, Control Over-eating, Binge Eating and Purging, Emotional Eating, Exercise Patterns and Attitudes). (baseline, post, 1-month post)
Yale Food Addiction Scale | 5 months
  The YFAS-c is a validated measure of addictive-like eating behavior based on the Diagnostic and Statistical Manual of Mental Disorder V diagnostic criteria for substance use disorders. (baseline, post, 1-month post)
International Physical Activity Questionnaire | 5 months
  The IPAQ is a seven item self-report questionnaire that asks how much time the participant has engaged in physical activity during the past seven days, including mild to vigorous activity. (baseline, post, 1-month post)
Nicotine use as measured by the CRAFFT section C | 5 months
  Nicotine use (vaping or other tobacco products) will be assessed using Part C of the CRAFFT; it will be modified to assess past 30-day use rather than past year (Mitchell, Kelly, Gryczynski, Myers, O'Grady, Kirk, & Schwartz, 2014). (baseline, post, 1-month post)

OTHER OUTCOMES:
Reach and Retention Rates | 4 months
  Participation rates; characteristics of participants vs. non-participants; attrition rates; enrollment rates based on recruitment source

CONTACTS AND LOCATIONS:
Overall Officials: Vibha Singhal, MD, MBBS, MPH, Principal Investigator — University of California, Los Angeles
Locations (1):
- UCLA Marion Davies Children's Center, Los Angeles, California, United States